CLINICAL TRIAL: NCT07349927
Title: Impact of Parental Training in Endocrine Disruptors on the Excretion of Urinary Biomarkers of Exposure: a Randomised Controlled Pilot Study With Two Parallel Arms
Brief Title: Impact of Parental Training in Endocrine Disruptors on the Excretion of Urinary Biomarkers in Newborns
Acronym: FLOCON
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL24_0017; 2025-A01198-41 (Other: ID-RCB)
Record Dates: First submitted 2025-12-24; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Endocrine Disruptors in Newborns and Infants
Keywords: Endocrine Disruptors; Phtalate; Newborns; Exposition; Urinary biomarkers; Parental training
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at Month 1 either in the Training group or in the Control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Parents attending a training course on endocrine disruptors one month after enrolment (Month 1)
  Interventions: Behavioral: Training; Other: Questionnaires; Biological: Urinary dosage
- Control group (Other): Parents attending a training course on endocrine disruptors two months after enrolment (Month 2)
  Interventions: Behavioral: Training; Other: Questionnaires; Biological: Urinary dosage

INTERVENTIONS:
Behavioral: Training — Short 4-minute information video on EDs (the investigator present on site during the visit will provide additional information and answer any questions families may have) and a printed brochure (including a list of simple actions to take and reference websites to consult).
Other: Questionnaires — Knowledge and representation questionnaires around EDs Exposure questionnaires Behavior questionnaire HLS-EU16 questionnaire Satisfaction questionnaire
Biological: Urinary dosage — Urinary phtalates dosage

SUMMARY:
The impact of the environment on health, responsible for a quarter of all deaths worldwide and costing more than €160 billion a year, is difficult to assess because of the complexity of exposure and interactions. Endocrine disrupters (EDs), which are omnipresent in our daily lives, affect hormone metabolism and can have long-term consequences, including effects on subsequent generations. Although complete avoidance is impossible, it is possible to reduce exposure through simple measures.

EDs can be divided into two groups: those with a short half-life, which are rapidly eliminated through the urine, and those with a long half-life, such as PFAS (Per- and polyfluoroalkyl substances), which accumulate in the body. Short-half-life EPs are particularly interesting for interventional studies, as their rapid elimination means that the impact of actions can be measured in a few days.

Policies to combat EDs, such as phthalate-free cities, have been put in place, but impact assessments are still needed. The national plan to combat EDs is based on improving public knowledge, collecting data on impregnation and looking for alternatives.

Studies show that modifying diet and personal care products can reduce concentrations of ED biomarkers, but the results are difficult to transpose to France. The 'first 1,000 days' (pregnancy, birth, infancy) are a window of vulnerability, providing an ideal opportunity to provide information and reduce exposure.

Environmental health research focuses on assessing exposure using biomarkers and informing the public. Studies on newborns and infants, which are still rare, are essential for a better understanding of the risks. Interventions to limit exposure to EDs with short half-lives can have rapidly measurable effects, and randomised studies are needed to test these reduction strategies.

The hypothesis of the study is that practical parental training in simple gestures can reduce the urinary excretion of short-half-life EDs in infants.

This study will therefore provide data on the exposure of infants prior to dietary diversification and assess the impact of parental information on urinary ED levels.

ELIGIBILITY:
Inclusion Criteria:

* Newborns born at the Bron hospital after 37 weeks of amenorrhea
* Eutrophic
* Affiliated to a social security scheme or beneficiary of a similar scheme
* Consent signed by parents

Exclusion Criteria:

* Congenital anomaly diagnosed antenatally or postnatally
* Parents who do not speak French

Ages: 0 Days to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of the variation in urinary Mono-n-butyl-phthalate (MBP) levels in infants in the 'training' group versus the 'control' group between Month 1 and Month 2 | Month 1, Month 2
  Comparison of the variation in urinary Mono-n-butyl-phthalate (MBP) levels in infants in the 'training' group versus the 'control' group between Month 1 and Month 2

SECONDARY OUTCOMES:
Relative variation, between Month 1 and Month 2, in the 'training' group (parents trained at Month 1) compared to the 'control' group, in urinary concentrations of : Mono(2-ethyl-5-oxohexyl)-phthalate also called 5-oxo-MEHP | Month 1, Month 2
  Relative variation, between Month 1 and Month 2, in the 'training' group (parents trained at M1) compared to the 'control' group, in urinary concentrations of : Mono(2-ethyl-5-oxohexyl)-phthalate also called 5-oxo-MEHP
Relative variation, between Month 1 and Month 2, in the 'training' group (parents trained at Month 1) compared to the 'control' group, in urinary concentrations of Mono(2-ethyl-5-hydroxyhexyl)-phthalate also called 5-OH-MEHP | Month 1, Month 2
  Relative variation, between Month 1 and Month 2, in the 'training' group (parents trained at Month 1) compared to the 'control' group, in urinary concentrations of Mono(2-ethyl-5-hydroxyhexyl)-phthalate also called 5-OH-MEHP
Relative variation between Month 1 and Month 2 in the 'training' group (parent training at Month 1) compared with the 'control' group, in urinary concentration of Mono(5-carboxy-2-ethylpentyl)-phthalate also called 5-cx-MEPP | Month 1, Month 2
  Relative variation between Month 1 and Month 2 in the 'training' group (parent training at Month 1) compared with the 'control' group, in urinary concentration of Mono(5-carboxy-2-ethylpentyl)-phthalate also called 5-cx-MEPP
Relative variation, between Month 1 and Month 2, in the 'training' group (training of parents at Month 1) compared to the 'control' group, in urinary concentrations of Mono[2-(carboxymethyl)hexyl]-phthalate also called 2-cx-MMHP | Month 1, Month 2
  Relative variation, between Month 1 and Month 2, in the 'training' group (training of parents at Month 1) compared to the 'control' group, in urinary concentrations of Mono[2-(carboxymethyl)hexyl]-phthalate also called 2-cx-MMHP

CONTACTS AND LOCATIONS:
Locations (1):
- Service de gynécologie obstétrique, Hôpital Femme-Mère-Enfant, Bron, France